CLINICAL TRIAL: NCT00519181
Title: Open Label Study of the Clinical and Laboratory Effects of Valproic Acid In HAM/TSP
Brief Title: Safety and Efficiency Study of Valproic Acid In HAM/TSP
Acronym: VALPROHAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Pierre Zobda-Quitman (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-SO-2006-17
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2007-08-22 (Estimated); Status verified 2007-08

CONDITIONS: HTLV-I-Associated Myelopathy
Keywords: HTLV; HAM/TSP; VALPROIC ACID; PROVIRAL LOAD
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Valproic Acid — Valproic acid by oral route (20mg/Kg/day) during one year.

SUMMARY:
Reversible acetylation of the histone tails plays an important role in the control of specific gene expression. Mounting evidence has established that histone deacetylase inhibitors such as Valproic Acid (VPA)selectively induce cellular differentiation and apoptosis in variety of cancer cells. In a single-center, one year open-label trial, 19 HAM/TSP patients were treated with oral doses of VPA (20mg/Kg/day). Primary end-points were the therapeutic safety and the effect on HTLV-1 proviral load (a significant and sustained decrease was expected). Secondary end-point was the neurological status before and after one-year treatment.

ELIGIBILITY:
Inclusion Criteria:

* HAM/TSP patients diagnosed on WHO criteria
* Obtained informed consent.

Exclusion Criteria:

* Patients with hepatic or nephrologic disease
* Valproic Acid allergy
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Clinical and laboratory safety of Valproic Acid in HAM/TSP. Effect on HTLV-1 proviral load in peripheral blood mononuclear cells. | one year

SECONDARY OUTCOMES:
Neurological outcome. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephane OLINDO, MD, Principal Investigator — University Hospital Pierre Zobda-Quitman, Fort de France

REFERENCES:
- [Derived] Lezin A, Gillet N, Olindo S, Signate A, Grandvaux N, Verlaeten O, Belrose G, de Carvalho Bittencourt M, Hiscott J, Asquith B, Burny A, Smadja D, Cesaire R, Willems L. Histone deacetylase mediated transcriptional activation reduces proviral loads in HTLV-1 associated myelopathy/tropical spastic paraparesis patients. Blood. 2007 Nov 15;110(10):3722-8. doi: 10.1182/blood-2007-04-085076. Epub 2007 Aug 23. PMID 17717136